CLINICAL TRIAL: NCT06496997
Title: A Comparative Study of Glucocorticoids Efficacy in Acute Respiratory Distress Syndrome
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mahmoud Ezzat Musa Abdel Tawab, Teaching assistant in Clinical Pharmacy Department-Faculty of Pharmacy-Fayoum University, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Steroids Efficacy in ARDS
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Methylprednisolone; Dexamethasone; Hydrocortisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): 100 ARDS patients
  Interventions: Drug: Methylprednisolone
- Group 2 (Experimental): 100 ARDS patients
  Interventions: Drug: Dexamethasone
- Group 3 (Experimental): 100 ARDS patients
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Methylprednisolone — Methylprednisolone at a dose of 1 mg/kg/day (an average dose of 70 mg/day based on 70 kg body weight)
  Arms: Group 1
Drug: Dexamethasone — Dexamethasone at an equivalent dose of 13 mg/day
  Arms: Group 2
Drug: Hydrocortisone — Hydrocortisone at an equivalent dose of 350 mg/day
  Arms: Group 3

SUMMARY:
The aim of the work is to compare the efficacy of equivalent doses of methylprednisolone, dexamethasone and hydrocortisone in patients with ARDS

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is a secondary disease that follows-usually within 6-48 h-a primary disease of multifactorial etiology (most frequently pneumonia and extrapulmonary sepsis) associated with severe systemic inflammation. Inflammatory mediators released into the systemic circulation (systemic inflammation) from the site of infection reach the broad pulmonary capillary surface, producing severe and diffuse inflammatory exudate of the pulmonary lobules and resulting in hypoxemic respiratory failure.

In ARDS, systemic inflammation is activated by the nuclear factor-κB (NF-κB) signaling system and downregulated by activated glucocorticoid receptor α (GRα). In these patients, inadequate (endogenous glucocorticoid-activated) GRα-mediated downregulation of proinflammatory transcription factor NF-κB in circulating and tissue cells leads to higher initial levels and persistent elevation over time of plasma and bronchoalveolar lavage markers of inflammation, hemostasis, and tissue repair. Inadequate intracellular GRα-mediated anti-inflammatory activity for the severity of the patient's illness was recently termed critical illness-related corticosteroid insufficiency (CIRCI). Experimental and clinical research shows that CIRCI can be improved with quantitatively and temporally adequate glucocorticoid administration.

Glucocorticoids are commonly used in patients with acute respiratory distress syndrome (ARDS) or at-risk for ARDS with proposed mechanisms including reduction of local lung inflammation and dampening of systemic immune responses.

Clinical trials of glucocorticoids in patients with ARDS or at-risk from a pulmonary infection have had mixed results with some studies suggesting benefit and others showing no beneficial effects. Notably, the glucocorticoid agent, dose, and duration has varied widely between studies increasing the challenge of interpreting discordant findings.

In animal models of ARDS, glucocorticoids decreased the expression of pro-inflammatory mediators in lung tissue, including TNF-a, IL-1a, IL-1b, IL-6 and IL-12 p40, and reduces lung injury through the reduction of oxygen radicals produced by neutrophils. Beyond their anti-inflammatory effects during the acute phase of inflammation, glucocorticoids also contributed to the resolution of inflammation, trough reprogramming effects on macrophages.

Glucocorticoids have been administered during two distinct phases of ARDS, during the early stage of ARDS when inflammation is expected to be most important and during late phase of ARDS, when lung fibrosis predominates. The biological and pathological characteristics of these two entities differ greatly, explaining the observed conflicting results in the effects of glucocorticoids in these two distinct conditions.

The early phase of ARDS is characterized by major alveolar inflammation. Thus, glucocorticoids, potent anti-inflammatory agents, are theoretically expected to be relevant treatment for ARDS.

Late-stage ARDS is characterized histologically by ongoing inflammation with fibroproliferation, presence of hyaline membranes, and persistent diffuse alveolar damage, leading to prolonged mechanical ventilation and a higher risk of death. The largest multicenter placebo-controlled trial, found no evidence for beneficial effects of glucocorticoids initiated for late-stage ARDS.

ELIGIBILITY:
Inclusion Criteria:

We include patients receiving mechanical ventilation for hypoxemic respiratory failure if they met the diagnostic criteria for ARDS according to the American-European Consensus definition, as later reclassified on the basis of the 2012 Berlin criteria for the diagnosis of ARDS, defined as:

1. Presence of acute hypoxemic respiratory failure (an arterial oxygen partial pressure to fraction of inspired oxygen ratio (PaO2/FiO2) of ≤ 300 mm Hg, requiring supplemental oxygen administrated by simple face mask, nasal cannula, or other similar oxygen-delivery device to maintain oxygen saturation at greater than 93% within the first 48 h of the onset of ARDS)
2. Onset within 7 days of insult, or new (within 7 days) or worsening respiratory symptoms
3. Bilateral opacities on chest x-ray or CT not fully explained by effusions, lobar or lung collapse, or nodules
4. Cardiac failure not the primary cause of acute respiratory failure

Exclusion Criteria:

We exclude patients with acute hypoxemic respiratory failure caused by congestive heart failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
28-day mortality after enrolment | From enrollment to the end of treatment at 28 days

SECONDARY OUTCOMES:
The number of patients needing invasive mechanical ventilation | From enrollment to the end of treatment at 28 days
The Number of ventilator-free days | From enrollment to the end of treatment at 28 days
Duration of the ICU stay | From enrollment to the end of treatment at 28 days
Duration of hospitalization | From enrollment to the end of treatment at 28 days
Incidence of serious adverse events, including secondary infections, hyperglycemia, clinically important gastrointestinal bleeding, and hypertension | From enrollment to the end of treatment at 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Ezzat Elkmash, Teaching Assistant, Principal Investigator — Faculty of Pharmacy - Fayoum University; Raghda Roshdy Hussein, Assistant Professor, Study Director — Faculty of Pharmacy - Beni Suef University; Marwa Kamal Tolba, Assistant Professor, Study Director — Faculty of Pharmacy - Fayoum University; Marian Sobhi Saeed, Lecturer, Study Director — Faculty of Pharmacy - Beni Suef University; Mona Ibrahim Ahmed, Lecturer, Study Director — Faculty of Medicine - Fayoum University
Locations (1):
- Fayoum University, Al Fayyum, Egypt